CLINICAL TRIAL: NCT01145404
Title: Lapatinib Versus Lapatinib With Capecitabine as Second-line Treatment in Her2-Overexpressing Metastatic Gastro-Esophageal Cancer: A Randomized Phase II Trial
Brief Title: Trial of Lapatinib Versus Lapatinib With Capecitabine in Her2+ Metastatic Gastro-Esophageal Cancer
Acronym: GastroLap
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes of SoC for third line therapy resulting in poor recruitment
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2008-11-01-1015
Record Dates: First submitted 2010-05-21; First posted 2010-06-16 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: GastroEsophageal Cancer
Keywords: Her2 Gastro Gastric Esophageal Cancer
MeSH Terms: interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Lapatinib (Experimental): Lapatinib (Tyverb) po 1500mg daily d1-21, new cycle will be started on day 22 until progression.
  Interventions: Drug: Lapatinib
- Arm B (Experimental): Lapatinib po 1250mg daily d1-21; new cycle will be started on day 22 until progression
  Interventions: Drug: Lapatinib plus capecitabine

INTERVENTIONS:
Drug: Lapatinib — Lapatinib (Tyverb) po 1500mg daily d1-21, new cycle will be started on day 22 until progression.
  Other Names: Tyverb
  Arms: Arm A: Lapatinib
Drug: Lapatinib plus capecitabine — Lapatinib po 1250mg daily d1-21; new cycle will be started on day 22 until progression
  Other Names: Tyverb, Xeloda
  Arms: Arm B

SUMMARY:
Combining Erb inhibitors, such lapatinib, and TS inhibitors, such as capecitabine, may be a beneficial contribution to current treatment paradigms since preclinical data suggest that lapatinib alone can decrease TS mRNA and is synergistic with capecitabine in some cell lines, which may contribute to clinical benefit. The study described in this protocol has been designed to establish the anti-tumor activity of Lapatinib with or without capecitabine in the treatment of Her2 overexpressing metastatic gastric- and gastro-esophageal cancer, and to search for molecular correlates that may be associated with response to this compound.

The majority of patients with metastatic gastric and gastro-esophageal cancer undergo first-line combined chemotherapy (e.g. platin derivates and fluoropyrimidines, sometimes combined to a taxane), but the role of second-line chemotherapy has not yet been defined. Therefore, progression during or shortly after first-line chemotherapy is a medical condition no standard medical approach exists. The overexpression of EGFR and Her2 in gastric and gastroesophageal cancer make these indications prime candidate for treatment with the dual ErbB1/2 tyrosine kinase inhibitor (TKI) Lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach, including adenocarcinoma of the gastroesophageal junction and esophagus
* Metastatic disease
* Measurable disease (according to RECIST criteria)
* At least one prior chemotherapy for metastatic disease with progression during or no later than 6 months after last administration of chemotherapy. Chemotherapy must have contained a platinum compound (cisplatin or oxaliplatin)
* Her2 overexpression measured by FISH (amplification or increased gene copy number). Immunohistochemistry (ICH) 3+ can be included in case of an uncertain FISH test.
* Patient willing to allow for biomarker analyses on his tumor tissue.
* Written informed consent given prior to any protocol specific procedures according to the local regulatory requirements
* Age >= 18 years
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) <= 2
* Life expectancy > 3 months
* Adequate hematological, hepatic and renal function defined by: Hematology: Neutrophils >1.5x109/L; Platelets >100x109/L; Hemoglobin >8g/dL Hepatic function: Total bilirubin <=1.5xULN; ASAT (SGOT) and ALAT (SGPT) <= 2.5xULN; Alkaline phosphatase <5xULN. Renal function: The calculated creatinine clearance should be .60 mL/min
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib will be determined following review of their use by the local Principal Investigator. A list of medications and substances known or with the potential to interact with CYP450 isoenzymes is provided in: Cytochrome P-450 Enzymes and Drug metabolism. In: Lacy CF, Armstrong LL, Goldman MP, Lance LL eds. Drug Information Handbook 8TH ed. Hudson, OH; LexiComp Inc. 2000: 1364-1371
* Able to swallow and retain oral medication
* Negative pregnancy test (urine or serum) within 28 days prior to randomization for all women of childbearing potential (has to be verified within 7 days prior to randomization and during the study according the judgement of the investigator)
* Willingness to perform double-barrier contraception during study and 6 months after end of treatment
* Ability to understand and the willingness to sign a written informed consent document
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Previous non curatively treated malignant disease other than the current gastroesophageal cancer with a disease-free survival of less than 5 years
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
* History of active Hepatitis B or C or history of an HIV infection
* Active uncontrolled infection
* Treatment within any other clinical trial parallel to the treatment phase of the current study within 30 days prior to randomisation.
* Concurrent treatment with any other anti-cancer drug. Presence of other medication that may interfere with study treatment or the action of the investigational product or confuse the assessment of study results
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or to any excipients
* History of allergic reactions attributed to compounds of similar chemical composition to capecitabine, fluorouracil or to any excipients
* Known DPD deficiency
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors
* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Active cardiac disease, defined as:

  * History of uncontrolled or symptomatic angina
  * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation

    * Myocardial infarction < 6 months from randomization
    * Uncontrolled or symptomatic congestive heart failure (> New York Heart Association score 2)
    * Ejection fraction below the institutional normal limit
    * Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | about 10 month (until progression)
  Objective response rate (ORR, complete and partial remission according to RECIST criteria
  - all to be confirmed by at least two consecutive tumor response assessments within no shorter than 4 weeks)

SECONDARY OUTCOMES:
Time to tumor progression | about 10 month (until tumor progression)
  Time to tumor progression
Overall survival | about 16 month (6 month after progression)
  Overall survival
Safety and tolerability of study treatment (for parameters see description) | about 10 month (until progression)
  recording of AEs/SAEs, vital signs, ECG, LVEF, physical exams, lab values
Biomarker analysis | 1 month (during screening period)
  the definition of biomarkers that are associated with response or resistance to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, MD, Study Director — Academic Teaching Hospital Braunschweig
Locations (16):
- Germany (16):
  - CHARITÉ CAMPUS, VIRCHOW-KLINIKUM, UNIVERSITÄTSMEDIZIN BERLIN, Centrum 14, Medizinische Klinik mit Schwerpunkt Hämatologie und Onkologie, Berlin
  - Evangelisches Krankenhaus Bielefeld gGmbH, Klinik für Innere Medizin, Hämatologie/Onkologie und Palliativmedizin, Bielefeld
  - Medizinische Uniklinik, Knappschaftskrankenhaus Bochum, Bochum
  - Evangelische Kliniken Bonn gGmbH, Johanniter-Krankenhaus, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Kliniken Essen Mitte, Department of Medical Oncology and Hematology, Essen
  - Klinikum Esslingen, Klinik für Allgemeine Innere Medizin, Onkologie und Gastroenterologie, Esslingen am Neckar
  - Krankenhaus Nord West, Frankfurt
  - Universitätsklinikum Halle, Klinik für Innere Medizin IV, Halle
  - OncoResearch Lerchenfeld UG, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie, Endokrinologie, Hanover
  - NCT Heidelberg, Heidelberg
  - I. Med. Klinik und Poliklinik, Universitätsmedizin der Johannes Gutenberg-Universität, Mainz
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Klinikum rechts der Isar, München
  - Klinikum Regensburg, Klinik und Poliklinik für Innere Medizin I, Regensburg

REFERENCES:
- [Derived] Lorenzen S, Riera Knorrenschild J, Haag GM, Pohl M, Thuss-Patience P, Bassermann F, Helbig U, Weissinger F, Schnoy E, Becker K, Stocker G, Ruschoff J, Eisenmenger A, Karapanagiotou-Schenkel I, Lordick F. Lapatinib versus lapatinib plus capecitabine as second-line treatment in human epidermal growth factor receptor 2-amplified metastatic gastro-oesophageal cancer: a randomised phase II trial of the Arbeitsgemeinschaft Internistische Onkologie. Eur J Cancer. 2015 Mar;51(5):569-76. doi: 10.1016/j.ejca.2015.01.059. Epub 2015 Feb 16. PMID 25694417